CLINICAL TRIAL: NCT06490731
Title: Effects of Dexmedetomidine Versus Ketamine on Inflammatory Response and Hemodynamic in Patients With Intraabdominal Sepsis: A Randomized Controlled Study
Brief Title: Effects of Dexmedetomidine Versus Ketamine on Inflammatory Response and Hemodynamic in Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Ismail Abdelsabour, lecture of anesthesia and ICU, New Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: New valley anesthesia 4
Record Dates: First submitted 2024-06-20; First posted 2024-07-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-11

CONDITIONS: Haemodynamic Rebound
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients will receive dexmedetomidine (Active Comparator): Patients will receive dexmedetomidine (Precedex®; 200 µg/2 ml; at one µg/kg loading dose over 10 minutes followed by a 0.5 µg/kg/hr. maintenance dose for 48 hours Dexmedetomidine will be diluted in normal saline at a 4 µg/ ml concentration
  Interventions: Drug: Dexmedetomidine
- Patients will receive ketamine (Active Comparator): Patients will receive ketamine at one mg/kg IV loading dose over 10 minutes, then a continuous infusion starting at 300 µg /kg/hr over 48 hours
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive dexmedetomidine
  Arms: Patients will receive dexmedetomidine
Drug: Ketamine — patients Will receive ketamine
  Arms: Patients will receive ketamine

SUMMARY:
Inflammatory response and hemodynamic response in patients with intraabdominal sepsis and Effects of Dexmedetomidine versus ketamine on it .

DETAILED DESCRIPTION:
Severe sepsis is a major healthcare problem with a reported incidence of 1-2% in all hospitalizations. It is a major cause of death in intensive care units worldwide and is the second leading cause of death in noncoronary intensive care unit patients. Mortality remains high at 30-50% despite a better understanding of sepsis pathophysiology and improved advanced care in the past decade . It is defined as a life-threatening organ dysfunction with a Sequential Organ Failure Assessment (SOFA) score > 2 and a mortality of over 10% in hospitals . These patients suffer from circulatory disorders including decreased intravascular volume, peripheral vasodilatation, and myocardial dysfunction, increased metabolism, which may result in hypoxia due to the imbalance between systemic oxygen delivery and oxygen demand .

The pathophysiology of septic shock is well known. However, septic shock therapy is still limited, and the mortality of patients with septic shock remains high. The innate immune system is the first line of defense mechanism against pathogens . The activation of the immunocompetent cells, including macrophages, monocytes, natural killer cells, dendritic cells, and endothelial cells mediate the innate immune response to respond to pathogens or their components . Activated immune cells also secrete pro-inflammatory mediators such as cytokines interleukin (IL-1, IL-6, IL-8), tumor necrosis factor-α (TNF-α), prostaglandins, and histamine . These mediators act on vascular endothelial cells and cause vasodilation, increased vascular permeability, and recruitment of neutrophils to the tissue .

The coagulation cascade is activated locally by upregulating endothelial tissue factors and decreased thrombomodulin and its antithrombotic products .

Ketamine is one of the most rational anaesthetic and sedative agents for patients with sepsis because of its ability to maintain hemodynamics Ketamine also suppresses pro-inflammatory cytokines, apoptosis, and increases intracellular calcium . In the hyperinflammatory phase, ketamine can also reduce anti-inflammatory cytokines such as IL-10 in the hypoinflammatory phase. Ketamine was thought to reduce the risk of secondary infection in the hypoinflammatory phase. However, there has yet to be further research on this hypothesis . Therefore, ketamine is expected to be developed as a candidate for immunotherapy in sepsis.

Dexmedetomidine (alpha2 receptor agonist) has anti-inflammatory and anti-bacterial effects, which are superior to those of gamma-aminobutyric acid agonists, such as benzodiazepines and propofol . Furthermore, it also reduces neuronal apoptosis high doses of central alpha-2-agonists like dexmedetomidine increase vasopressor responsiveness Moreover, even in non-septic patients, alpha-2-agonists are associated with lower vasopressor requirements, increased arterial blood pressure, and enhanced baroreceptor response .

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients admitted to ICU after ileus surgery (perforated viscus, infarcted bowel, strangulated hernia, anastomotic leakage, diverticulitis, and intestinal obstruction), and who will be expected to require postoperative sedation and ventilation.

  * Abdominal sepsis was determined as organ dysfunction with a substantial change in overall SOFA score (2) ≥ 2 points because of intra-abdominal sepsis.

Exclusion Criteria:

* • Known allergy to ketamine, dexmedetomidine,

  * Confirmed pregnancy,
  * Heart failure (class 3 or 4 of the New York Heart Association),
  * Renal failure (RIFLE classification),
  * Liver failure (manifested by serum total protein concentration <3 g/dl and total bilirubin >5 mg/dl)
  * Known or suspected brain death.
  * Patients who receive neuromuscular blockers during the first 48 hours of ICU admission will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 48 hours
  Effect of the study drugs as sedative agents on blood pressure in mechanically ventilated septic patients after abdominal exploration for intestinal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ismail Abdel Sabour, MD, Principal Investigator — NewValley University
Locations (1):
- asyut University, Asyut, Egypt